CLINICAL TRIAL: NCT01108965
Title: A Flow Monitor for Pediatric Hydrocephalic Shunts
Brief Title: Study of Shunt Flow Sensor Accuracy in Extra-ventricular Drains.
Status: Completed | Type: Observational
Sponsor: Transonic Systems Inc. (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: TSI-C-HYDRO-2A-H; 5R44NS049680-03 (NIH)
Record Dates: First submitted 2010-04-21; First posted 2010-04-22 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Hydrocephalus; Nervous System Diseases; Infant, Newborn Diseases
Keywords: Hydrocephalus; Shunt Dysfunction; Shunt Flow
MeSH Terms: conditions — Hydrocephalus; Nervous System Diseases; Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid samples are to be retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Extraventricular Drainage: Includes hydrocephalus patients that are in recovery from shunt explanation.

SUMMARY:
The study hypothesis is that an ultrasonic flow sensor can accurately measure flow in hydrocephalic shunts.

The ultrasonic sensor will measure cerebrospinal fluid drainage in hydrocephalus patients with external ventriculostomies and extra-ventricular drainage systems. The sensor measurements will be compared with the volume of fluid collected by the drainage bag.

After a 24-hour measurement period, the doctor will change the drainage bag position to simulate the patient sitting up and leaning back, to see if this temporarily stops flow through the drainage line.

This data will show whether the sensor accurately measures typical drainage flows seen in hydrocephalus patients. This research will help develop an implantable flow monitor for pediatric hydrocephalus patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hydrocephalus
* Instrumented with an Extraventricular drainage system

Exclusion Criteria:

* Not diagnosed with hydrocephalus
* Not instrumented with an extraventricular drainage system

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hydrocephalus patients under the care of SUNY Upstate Medical University
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2010-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Volumetric flow of patient cerebrospinal fluid through an Extra-Ventricular Drainage system. | 24 hour-period

SECONDARY OUTCOMES:
Recording of the pressure waveform related to the volumetric flow of patient cerebrospinal fluid through an Extra-Ventricular Drainage system. | 24 hour period

CONTACTS AND LOCATIONS:
Overall Officials: Cornelis J Drost, Principal Investigator — Transonic Systems Inc.; Satish Krishnamurthy, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States